CLINICAL TRIAL: NCT02705963
Title: A Phase I, Open-Label Study to Determine the Effect of Repeat Dosing of Trametinib on the Pharmacokinetics of a Combined Oral Contraceptive (Norethindrone Plus Ethinyl Estradiol) in Female Patients With Solid Tumors
Brief Title: A Drug-Drug Interaction Study to Assess the Effect of Trametinib on the Pharmacokinetics of an Oral Contraceptive in Female Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMT212X2102
Record Dates: First submitted 2016-02-22; First posted 2016-03-11 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2021-10

CONDITIONS: Solid Tumors
MeSH Terms: interventions — trametinib; Contraceptives, Oral; Norethindrone; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Contraceptive / Trametinib (Experimental): In treatment period 1 of the PK Phase patients will take the Oral Contraceptive once daily from Days 1-5. Period 2 of the PK Phase starts on Day 6 when patients take both the Oral Contraceptive and trametinib once daily from Days 6 to 21. Patients may continue dosing with trametinib only once daily from Day 22 onwards (post PK Phase).
  Interventions: Drug: Trametinib; Drug: Oral Contraceptive (1mg norethindrone, 0.035mg ethinyl estradiol)

INTERVENTIONS:
Drug: Trametinib — Each tablet is 2mg trametinib to be taken orally once daily.
Drug: Trametinib — Each tablet is 0.5mg trametinib to be taken orally once daily. 0.5mg tablets may be used if a dose reduction is required.
Drug: Oral Contraceptive (1mg norethindrone, 0.035mg ethinyl estradiol) — Combined oral contraceptive to be taken orally once daily.

SUMMARY:
The purpose of this study is to evaluate the effect of trametinib once daily on the pharmacokinetics (PK) of a daily dosing oral contraceptives (OCs) containing norethindrone (NE) and ethinyl estradiol (EE) in female patients with solid tumors. The PK of trametinib and its metabolite M5 will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of a solid tumor malignancy (except for any excluded malignancies listed in the Exclusion Criteria) that is not responsive to standard therapy(ies) or for which there is no approved therapy.
* Meets one of the following criteria: Is currently on a stable regimen of an oral contraceptive containing 1mg NE and 0.035mg EE, or Is willing to switch to a regimen of an oral contraceptive containing 1mg NE and 0.035mg EE from a stable regimen of an alternate OC, or Is willing to start a regimen of an oral contraceptive containing 1mg NE and 0.035mg EE.
* Meets one of the following criteria: Is post-menopausal, or, Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during dosing and for four months after stopping medication.
* Has no prior treatment-related toxicities >Grade 1 (except alopecia) at the time of enrolment.
* Patient must meet the following laboratory values at the screening visit: Absolute Neutrophil Count ≥1.5 x 109/L. Platelets ≥75 x 109/L. Hemoglobin (Hgb) ≥9 g/dL. Serum creatinine <1.5 mg/dL. Total bilirubin ≤1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). Aspartate transaminase (AST) ≤ 3.0 x ULN, except for patients with liver metastasis, who may only be included if AST ≤5.0 x ULN. Alanine transaminase (ALT) ≤ 3.0 x ULN, except for patients with liver metastasis or tumor infiltration, who may only be included if ALT ≤5.0 x ULN. Prothrombin time (PT)/International normalized ratio (INR) and Partial thromboplastin time (PTT) ≤1.5xULN. Note: patients receiving therapeutic anticoagulation agents prior screening are permitted. Albumin 2.5 g/dL.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

Exclusion Criteria:

* History or current diagnosis of cardiac disease indicating significant risk of safety for patients participating in the study such as uncontrolled or significant cardiac disease
* Has had any major surgery, extensive radiotherapy, or anti-cancer therapy (e.g., chemotherapy with delayed toxicity, biologic therapy, or immunotherapy) within 21 days prior to enrolment and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to enrolment. Prolonged immobilization must have resolved prior to enrolment.
* Has a known or suspected carcinoma that is excluded as administration of Oral Contraceptive would be contraindicated.
* Has a history of another malignancy.
* Has a history of interstitial lung disease or pneumonitis.
* Has a history of RVO.
* Has a history of any of conditions that would contraindicate administration of an OC
* Has symptomatic or untreated leptomeningeal, brain metastases, or spinal cord compression.

Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: AUCtau of NE and EE alone and in combination with trametinib | Day 5 and 6 and 21 and 22
  To evaluate the effect of multiple doses of trametinib (2 mg once daily) on the steady state pharmacokinetics of combination OC (NE and EE) in female patients with solid tumors.
Pharmacokinetics parameter: AUClast of NE and EE alone and in combination with trametinib | Day 5 and 6 and 21 and 22
  To evaluate the effect of multiple doses of trametinib (2 mg once daily) on the steady state pharmacokinetics of combination OC (NE and EE) in female patients with solid tumors.
Pharmacokinetics parameter: Cmax of NE and EE alone and in combination with trametinib | Day 5 and 6 and 21 and 22
  To evaluate the effect of multiple doses of trametinib (2 mg once daily) on the steady state pharmacokinetics of combination OC (NE and EE) in female patients with solid tumors.
Pharmacokinetics parameter: Tmax of NE and EE alone and incombination with trametinib | Days 5 and 6 and 21 and 22
  To evaluate the effect of multiple doses of trametinib (2 mg once daily) on the steady state pharmacokinetics of combination OC (NE and EE) in female patients with solid tumors.

SECONDARY OUTCOMES:
Pharmacokinetics parameter: AUClast of M5 | Day 21 and 22
  Characterize PK of metabolite M5
Pharmacokinetics parameter: AUCtau of M5 | Day 21 and 22
  Characterize PK of metabolite M5
Pharmacokinetics parameter: Cmax of M5 | Day 21 and 22
  Characterize PK of metabolite M5
Pharmacokinetics parameter: Tmax of M5 | Day 21 and 22
  Characterize PK of metabolite M5

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (2):
  - Karmanos Cancer Institute Karmanos Cancer Institute, Detroit, Michigan
  - University of Oklahoma, Oklahoma City, Oklahoma
- Belgium (2):
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Namur
- Novartis Investigative Site, Maastricht, Netherlands
- Novartis Investigative Site, Málaga, Spain
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- See also: Results for CTMT212X2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17699
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=612